CLINICAL TRIAL: NCT00421707
Title: A Phase 2 PoC in IBS Patients With the CRF1 Receptor Anatgonist, GSK876008
Brief Title: Randomized Placebo Controlled Efficacy And Safety Study Investigating GW876008 In Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CRI105626
Record Dates: First submitted 2007-01-10; First posted 2007-01-12 (Estimated); Results first posted 2017-12-26 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2017-11

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: Irritable Bowel Syndrome safety
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — GW 876008

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GW876008 (Experimental): GW876008
  Interventions: Drug: GW876008
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: GW876008; Other: Placebo

INTERVENTIONS:
Drug: GW876008
Other: Placebo
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled, randomised crossover study to investigate the efficacy and safety of GW876008

ELIGIBILITY:
Inclusion Criteria:

* The subject has been diagnosed with IBS consistent with the Rome II Criteria as adapted in Appendix 3 of the protocol
* The subject has normal results from a flexible sigmoidoscopy, colonoscopy, or a flexible sigmoidoscopy plus barium enema, according to subject's age, within 5 years of randomization. Otherwise, the appropriate procedure(s) must be performed and normal results obtained during the 7-day procedure window (prior to randomization):

If the subject is < 50 years of age and has not had a colonic examination within 5 years of the Screening Visit, flexible sigmoidoscopy, or colonoscopy must be performed.

If the subject is = 50 years of age and has not had a colonic examination within 5 years of the Screening Visit, a colonoscopy or flexible sigmoidoscopy plus barium enema must be performed.

* Colonic procedure results must be known prior to randomization into the study and dispensing study medication
* During the two-week screening phase, the subject must have conducted self assessments on = 10 days of 14 day (with 80% compliance on daily IVRS calls) compliance assessment using the telephone data entry system

Exclusion Criteria:

* As a result of any of the medical interview, physical examination, evaluation of mental state and psychiatric history or screening investigations the physician
* Subject reported no stool for 7 consecutive days during the two-week screening phase responsible considers the subject unfit for the study
* The subject has a concurrent illness or disability that may affect the interpretation of clinical data, or otherwise contraindicates participation in this clinical study (e.g., an unstable cardiovascular, autoimmune, renal, hepatic, pulmonary, endocrine, metabolic, gastrointestinal, haematological, or neurological condition).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2006-10-14 (Actual); Primary Completion 2008-06-25 (Actual); Study Completion 2008-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- United States (17):
  - GSK Investigational Site, Sherwood, Arkansas
  - GSK Investigational Site, Concord, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Monroe, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Lynchburg, Virginia
- Canada (3):
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Saskatoon, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 132 participants with irritable bowel syndrome (IBS), as classified by the Rome II criteria for IBS, but otherwise healthy, were randomized in this study. Study was conducted at 20 centers (14 centers in united states, six centers in Canada) from 14 October 2006 to 25 June 2008
Groups:
- Sequence A/X/B: As per the treatment sequence A/X/B, during period 1, eligible participants received GW876008 125 milligram (mg) (A) (1 x GW876008 100 mg and 1 x GW876008 25 mg ) once daily for 6 weeks, followed by a washout period (X) of 3 weeks where participants received matching placebo once daily followed by period 2 where participants received matching placebo (B) once daily for 6 weeks. Participants were instructed to take 1 tablet from each of the 2 bottles; 25 mg and 100 mg (specific for that dispensing period) orally in the morning with food. At the day of the Weeks 3, 6, 9, 12 and 15 Visit, participants were instructed not take their dose prior to their visit which was scheduled for the morning, they were instructed to take their dose at the site after collection of a pre-dose pharmacokinetic (PK) blood sample.
- Sequence B/X/A: As per the treatment sequence B/X/A, during period 1, eligible participants received matching placebo (B) once daily for 6 weeks followed by a washout period (X) of 3 weeks where participants received matching placebo once daily followed by period 2 where participants received GW876008 125 mg (A) (1 x GW876008 100 mg and 1 x GW876008 25 mg ) once daily for 6 weeks. Participants were instructed to take 1 tablet from each of the 2 bottles; 25 mg and 100 mg (specific for that dispensing period) orally in the morning with food. At the day of the Weeks 3, 6, 9, 12 and 15 Visit, participants were instructed not take their dose prior to their visit which was scheduled for the morning, they were instructed to take their dose at the site after collection of a pre-dose PK blood sample.
Period: Period 1: Treatment Period 1
Arm/Group | Sequence A/X/B | Sequence B/X/A
Started | 67 | 65
Completed | 56 | 56
Not Completed | 11 | 9
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Adverse Event | 7 | 2
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 1 | 0
Period: Period 2: Washout
Arm/Group | Sequence A/X/B | Sequence B/X/A
Started | 56 | 56
Completed | 55 | 52
Not Completed | 1 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other: Pregnancy | 0 | 1
Period: Period 3:Treatment Period 2
Arm/Group | Sequence A/X/B | Sequence B/X/A
Started | 55 | 52
Completed | 53 | 49
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Sequence A/X/B: As per the treatment sequence A/X/B, during period 1, eligible participants received GW876008 125 mg (A) (1 x GW876008 100 mg and 1 x GW876008 25 mg ) once daily for 6 weeks, followed by a washout period (X) of 3 weeks where participants received matching placebo once daily followed by period 2 where participants received matching placebo (B) once daily for 6 weeks. Participants were instructed to take 1 tablet from each of the 2 bottles; 25 mg and 100 mg (specific for that dispensing period) orally in the morning with food. At the day of the Weeks 3, 6, 9, 12 and 15 Visit, participants were instructed not take their dose prior to their visit which was scheduled for the morning, they were instructed to take their dose at the site after collection of a pre-dose pharmacokinetic (PK) blood sample.
- Total: Total of all reporting groups
Arm/Group | Sequence A/X/B | Sequence B/X/A | Total
Number analyzed (Participants) | 67 | 65 | 132
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.1 (11.74) | 43.0 (11.43) | 43.5 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 48 | 100
  Male | 15 | 17 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 58 | 52 | 110
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Average Adequate Relief Rate During the Last 4 Weeks of the Treatment Periods (Weeks 3-6. in Period 1, Weeks 12-15 in Period 2).
Description: For the assessment of average adequate relief rate from IBS symptoms for a participant was planned by collecting the response of a question 'In the past seven days have you had adequate relief of your IBS pain or discomfort? However, in error, the question was not collected in the IVRS system. Therefore, data for this endpoints was not collected during this study.
Time Frame: Up to Day 105 (weeks 3-6. in period 1, weeks 12-15 in period 2)
Population: Intent to Treat population comprised of all participants who were randomized to treatment, who received at least one dose of double blind medication and for whom at least one valid post baseline efficacy assessment was available.
Groups:
- GW876008 125 mg: Eligible participants received GW876008 125 mg once daily for 6 weeks. Participants were instructed to take 1 tablet from each of the 2 bottles; 25 mg and 100 mg orally in the morning with food. At the day of the Weeks 3, 6, 9, 12 and 15 Visit, participants were instructed not take their dose prior to their visit which was scheduled for the morning, they were instructed to take their dose at the site after collection of a pre-dose PK blood sample.
- Placebo: Eligible participants received matching placebo orally once daily for 6 weeks. Participants were instructed to take 1 tablet from each of the 2 bottles; 25 mg and 100 mg orally in the morning with food. At the day of the Weeks 3, 6, 9, 12 and 15 Visit, participants were instructed not take their dose prior to their visit which was scheduled for the morning, they were instructed to take their dose at the site after collection of a pre-dose PK blood sample.
- Placebo Washout: Eligible participants received washout placebo orally once daily for 3 weeks. Participants were instructed to take 1 tablet from each of the 2 bottles; 25 mg and 100 mg orally in the morning with food. At the day of the Weeks 3, 6, 9, 12 and 15 Visit, participants were instructed not take their dose prior to their visit which was scheduled for the morning, they were instructed to take their dose at the site after collection of a pre-dose PK blood sample.
Arm/Group | GW876008 125 mg | Placebo | Placebo Washout
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Changes in Weekly Adequate Relief Rates During the Treatment Periods (Weeks 1-6 in Period 1 and Weeks 9-15 in Period 2).
Description: For the assessment of changes in weekly adequate relief rates during the treatment periods was planned by collecting the response of a question. Overall response was defined as having achieved adequate relief in last 4 weeks. However, in error, the question was not collected in the IVRS system. Therefore, data for this endpoints was not collected during this study.
Time Frame: Up to Day 105 (weeks 1-6 in period 1 and weeks 9-15 in period 2).
Population: Intent to Treat population.
Arm/Group | GW876008 125 mg | Placebo | Placebo Washout
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Adequate Relief of IBS Pain and Discomfort on All 4 of the Last 4 Weeks of the Treatment Phase Treatment Periods 1 and 2
Description: For the assessment of average adequate relief rate from IBS symptoms for a participant was planned by collecting the response of a question whether weekly adequate relief from IBS symptoms was achieved?. However, in error, the question was not collected in the IVRS system. Therefore, data for this endpoints was not collected during this study.
Time Frame: Up to Day 105
Population: Intent to Treat population
Arm/Group | GW876008 125 mg | Placebo | Placebo Washout
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Mean Global Improvement Scale (GIS) Responder Rate Over the Last Four Weeks by Regimen
Description: The GIS is comprised of ten questions, all rated on a seven point scale ranging from substantially worse (7) to substantially improved (1). GIS assesses the participant's improvement (or worsening) as assessed by the clinician on a 7-point scale: 1: very much improved; 2: much improved; 3: minimally improved; 4: no change; 5: minimally worse; 6: much worse; or 7: very much worse for diarrhea, constipation, stool frequency, stool consistency, urgency, bloating, incomplete evacuation, and straining. Values reported are less than the minimum score on scale as the rate is the proportion of the last four weeks that the participant is a responder.
Time Frame: Up to Day 105 (weeks 3-6 in period 1, weeks 12-15 in period 2)
Population: Intent to Treat population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of participants responded
Arm/Group | GW876008 125 mg | Placebo
Number analyzed (Participants) | 117 | 117
Proportion of participants responded
  Pain and Discomfort | 0.26 (0.357) | 0.22 (0.334)
  diarrhea | 0.30 (0.377) | 0.28 (0.383)
  Constipation | 0.18 (0.319) | 0.16 (0.295)
  Stool Frequency | 0.25 (0.362) | 0.24 (0.349)
  Stool Consistency | 0.24 (0.370) | 0.21 (0.345)
  Urgency | 0.24 (0.365) | 0.25 (0.363)
  Bloating | 0.18 (0.329) | 0.16 (0.287)
  Incomplete Evacuation | 0.19 (0.350) | 0.16 (0.307)
  Straining | 0.19 (0.341) | 0.19 (0.319)
  IBS Symptoms | 0.32 (0.403) | 0.26 (0.357)

5. Primary Outcome: Ratings on Irritable Bowel Syndrome Quality of Life (IBSQoL) Scale
Description: The IBSQoL is a self-report quality-of-life measure specific to IBS that can be used to assess the impact of IBS and its treatment. The IBSQoL consists of 30 statements about bowel problems, which formed 9 scales: emotional health, mental health, health belief, sleep, energy, physical functioning, diet, social role, physical role and sexual relation. All 9 scales were rated on a five-point response scale ranging from 1 (always) to 5 (never). Scores for individual items were averaged to obtain a total score for each subscale of IBSQoL. Then transformed to a 0-100 scale for ease of interpretation with higher scores indicating better IBS-specific quality of life. Transformed scale score = (raw score - lowest possible scale score)/ (scale range) X 100. The data presented for individual scale.
Time Frame: Up to Day 105 (weeks 3-6 in period 1, weeks 12-15 in period 2)
Population: Intent to Treat population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | GW876008 125 mg | Placebo | Placebo Washout
Number analyzed (Participants) | 106 | 114 | 112
Score on a scale
  Emotional | 15.35 (3.852) | 15.72 (3.674) | 15.39 (3.595)
  Mental Health | 21.07 (4.141) | 21.39 (3.116) | 21.21 (3.253)
  Sleep | 12.49 (2.489) | 12.47 (2.570) | 12.79 (2.551)
  Energy | 8.22 (1.892) | 8.25 (1.986) | 8.21 (1.870)
  Physical Functioning: number analyzed (Participants) | 105 | 112 | 110
  Physical Functioning | 5.23 (1.683) | 5.63 (2.282) | 5.50 (2.067)
  Food/Diet | 14.27 (3.131) | 14.74 (2.894) | 14.60 (2.890)
  Social | 16.11 (3.783) | 16.39 (3.414) | 16.43 (3.767)
  Role-Physical | 15.16 (4.472) | 15.85 (4.189) | 15.44 (4.261)
  Sexual Relations: number analyzed (Participants) | 70 | 81 | 78
  Sexual Relations | 12.30 (3.122) | 13.10 (2.667) | 12.73 (3.056)

6. Secondary Outcome: Number of Participants With Improvements in Pain and Discomfort
Description: Number of participants with improvements in pain and discomfort on GIS were presented. GIS assesses the participant's improvement (or worsening) as assessed by the clinician on a 7-point scale: 1: very much improved; 2: much improved; 3: minimally improved; 4: no change; 5: minimally worse; 6: much worse; or 7: very much worse on specified time points. Responder = Yes if A responder answered either 'moderately improved' or 'substantially improved'.
Time Frame: Up to Day 105 (weeks 3-6 in period 1, weeks 12-15 in period 2)
Population: Intent to Treat population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GW876008 125 mg | Placebo | Placebo Washout
Number analyzed (Participants) | 117 | 119 | 112
Participants
  Week 1, Yes | 25 | 20 | 24
  Week 1, No | 92 | 95 | 85
  Week 2, Yes | 25 | 18 | 24
  Week 2, No | 92 | 98 | 88
  Week 3, Yes | 30 | 22 | 31
  Week 3, No | 87 | 96 | 81
  Week 4, Yes | 30 | 26 | 0
  Week 4, No | 87 | 91 | 0
  Week 5, Yes | 31 | 28 | 0
  Week 5, No | 86 | 89 | 0
  Week 6, Yes | 31 | 26 | 0
  Week 6, No | 86 | 91 | 0

7. Secondary Outcome: Change From Baseline in Pain Severity Scores
Description: Pain severity scores from the 11-point scale and it's corresponding change from Baseline scores was summarized by treatment group for the last 4 weeks (i.e. weeks 3-6 and Weeks 12-15) of treatment period. Scale from 0 to 10, 0 meaning no pain, 10 worst possible pain. Lower values represent a better outcome. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting baseline value from specified time point value. Reported data values are lesser than minimum score on scale as change from Baseline is reported.
Time Frame: Baseline (Day 1) and up to Day 105 (weeks 3-6 in period 1, weeks 12-15 in period 2)
Population: Intent to Treat population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | GW876008 125 mg | Placebo
Number analyzed (Participants) | 67 | 67
Score on a scale
  Stool consistency, Week 3-6 | -0.04 (0.654) | 0.03 (0.571)
  Stool frequency, Week 3-6 | -0.25 (0.905) | -0.35 (0.932)
  5 point pain severity, Week 3-6 | -0.89 (0.745) | -0.87 (0.753)
  IBS Symptoms, Week 3-6 | -0.58 (0.501) | -0.55 (0.498)
  Nausea severity, Week 3-6 | -0.27 (0.546) | -0.31 (0.525)
  Vomitting severity, Week 3-6 | -0.00 (0.072) | -0.02 (0.129)
  Burping severity, Week 3-6 | -0.36 (0.568) | -0.35 (0.599)
  Feeling full severity, Week 3-6 | -0.54 (0.729) | -0.49 (0.660)
  Feeling excessively full severity, Week 3-6 | -0.48 (0.726) | -0.48 (0.671)
  Bloating severity, Week 3-6 | -0.78 (0.798) | -0.77 (0.684)
  Diarrhoea severity, Week 3-6 | -0.43 (0.619) | -0.42 (0.573)
  Constipation severity, Week 3-6 | -0.31 (0.592) | -0.33 (0.546)
  Urgency severity, Week 3-6 | -0.58 (0.605) | -0.45 (0.617)
  Straining severity, Week 3-6 | -0.31 (0.568) | -0.34 (0.556)
  Incomplete evacuation severity, Week 3-6 | -0.47 (0.704) | -0.48 (0.587)
  Flatulence severity, Week 3-6 | -0.54 (0.632) | -0.50 (0.593)
  Heartburn severity, Week 3-6 | -0.18 (0.617) | -0.17 (0.544)

8. Secondary Outcome: Percentages of Pain-free Days
Description: Abdominal pain free days are those days where the participant reported a score of '0' for abdominal pain at its worst. Abdominal Pain (in the last 24 hours) is based on an 11-point scale where 0 represents no abdominal pain and 10 represents very severe abdominal pain.
Time Frame: Up to Day 105 (weeks 3-6 in period 1, weeks 12-15 in period 2)
Population: Intent to Treat population. Only those participants available at the specified time points were analyzed. Washout period was of 3 weeks only. Thus, these categories are not applicable for placebo washout arm.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | GW876008 125 mg | Placebo | Placebo Washout
Number analyzed (Participants) | 117 | 119 | 112
Percentage of days
  Week 1: number analyzed (Participants) | 117 | 116 | 111
  Week 1 | 27.25 (33.261) | 24.38 (31.015) | 34.92 (37.032)
  Week 2: number analyzed (Participants) | 117 | 119 | 111
  Week 2 | 32.72 (37.331) | 28.21 (34.768) | 32.82 (36.528)
  Week 3: number analyzed (Participants) | 115 | 118 | 111
  Week 3 | 38.14 (38.113) | 32.45 (36.870) | 35.14 (37.688)
  Week 4: number analyzed (Participants) | 113 | 117 | 0
  Week 4 | 35.52 (36.075) | 33.09 (38.059) |
  Week 5: number analyzed (Participants) | 111 | 115 | 0
  Week 5 | 36.04 (38.277) | 32.30 (35.303) |
  Week 6: number analyzed (Participants) | 109 | 115 | 0
  Week 6 | 39.97 (42.315) | 34.29 (37.358) |
  Week 3-6: number analyzed (Participants) | 117 | 119 | 0
  Week 3-6 | 36.87 (35.470) | 33.31 (32.875) |

9. Secondary Outcome: Number of Participants With Improvements in Bowel Function and Changes in Individual Bowel Symptoms/Function
Description: The GIS comprised of ten questions, all rated on a seven point scale ranging from substantially worse (7) to substantially improved (1). GIS assesses the participant's improvement (or worsening) as assessed by the clinician on a 7-point scale: 1: very much improved; 2: much improved; 3: minimally improved; 4: no change; 5: minimally worse; 6: much worse; or 7: very much worse. Number of participants who showed improvement and changes on the scale were presented. Participants were counted as "Yes" if they scored 1-3, and as "No" if they scored 4-7.
Time Frame: Up to Day 105 (weeks 3-6 in period 1, weeks 12-15 in period 2)
Population: Intent to Treat population.
Measure: Count of Participants; unit: Participants
Arm/Group | GW876008 125 mg | Placebo | Placebo Washout
Number analyzed (Participants) | 117 | 119 | 112
Participants
  Diarrhea, Week 1, Yes | 28 | 28 | 33
  Diarrhea, Week 1, No | 89 | 87 | 76
  Diarrhea,Week 2,Yes | 30 | 30 | 32
  Diarrhea, Week 2, No | 87 | 86 | 80
  Diarrhea, Week 3, Yes | 34 | 33 | 29
  Diarrhea, Week 3, No | 83 | 85 | 83
  Diarrhea, Week 4, Yes | 32 | 31 | 0
  Diarrhea, Week 4, No | 85 | 86 | 0
  Diarrhea, Week 5, Yes | 41 | 36 | 0
  Diarrhea, Week 5, No | 76 | 81 | 0
  Diarrhea, Week 6,Yes | 33 | 29 | 0
  Diarrhea, Week 6,No | 84 | 88 | 0
  Constipation, Week 1, Yes | 15 | 14 | 16
  Constipation, Week 1 ,No | 102 | 101 | 93
  Constipation, Week 2, Yes | 18 | 15 | 19
  Constipation, Week 2, No | 99 | 101 | 93
  Constipation, Week 3, Yes | 19 | 15 | 17
  Constipation, Week 3, No | 98 | 103 | 95
  Constipation, Week 4, Yes | 21 | 20 | 0
  Constipation, Week 4, No | 96 | 97 | 0
  Constipation, Week 5, Yes | 22 | 18 | 0
  Constipation, Week 5, No | 95 | 99 | 0
  Constipation, Week 6, Yes | 23 | 20 | 0
  Constipation, Week 6, No | 94 | 97 | 0
  Stool frequency, Week 1, Yes | 21 | 19 | 22
  Stool frequency, Week 1, No | 96 | 96 | 87
  Stool frequency, Week 2, Yes | 24 | 23 | 24
  Stool frequency, Week 2, No | 93 | 93 | 88
  Stool frequency, Week 3, Yes | 27 | 25 | 21
  Stool frequency, Week 3, No | 90 | 93 | 91
  Stool frequency, Week 4, Yes | 26 | 29 | 0
  Stool frequency, Week 4, No | 91 | 88 | 0
  Stool frequency, Week 5, Yes | 31 | 30 | 0
  Stool frequency, Week 5, No | 86 | 87 | 0
  Stool frequency, Week 6, Yes | 34 | 27 | 0
  Stool frequency, Week 6, No | 83 | 90 | 0
  Stool consistency, Week 1, Yes | 17 | 18 | 22
  Stool consistency, Week 1, No | 100 | 97 | 87
  Stool consistency, Week 2, Yes | 21 | 20 | 22
  Stool consistency, Week 2, No | 96 | 96 | 90
  Stool consistency, Week 3, Yes | 27 | 23 | 23
  Stool consistency, Week 3, No | 90 | 95 | 89
  Stool consistency, Week 4, Yes | 26 | 27 | 0
  Stool consistency, Week 4, No | 91 | 90 | 0
  Stool consistency, Week 5, Yes | 30 | 27 | 0
  Stool consistency, Week 5, No | 87 | 90 | 0
  Stool consistency, Week 6, Yes | 28 | 23 | 0
  Stool consistency, Week 6, No | 89 | 94 | 0
  Sense of urgency, Week 1, Yes | 24 | 17 | 22
  Sense of urgency, Week 1, No | 93 | 98 | 87
  Sense of urgency, Week 2, Yes | 24 | 26 | 27
  Sense of urgency, Week 2, No | 93 | 90 | 85
  Sense of urgency, Week 3, Yes | 30 | 31 | 24
  Sense of urgency, Week 3, No | 87 | 87 | 88
  Sense of urgency, Week 4, Yes | 28 | 28 | 0
  Sense of urgency, Week 4, No | 89 | 89 | 0
  Sense of urgency, Week 5, Yes | 27 | 29 | 0
  Sense of urgency, Week 5, No | 90 | 88 | 0
  Sense of urgency, Week 6, Yes | 29 | 28 | 0
  Sense of urgency, Week 6, No | 88 | 89 | 0
  Bloating, Week 1, Yes | 19 | 14 | 17
  Bloating, Week 1, No | 98 | 101 | 92
  Bloating, Week 2, Yes | 22 | 14 | 18
  Bloating, Week 2, No | 95 | 102 | 94
  Bloating, Week 3, Yes | 19 | 19 | 19
  Bloating, Week 3, No | 98 | 99 | 93
  Bloating, Week 4, Yes | 23 | 20 | 0
  Bloating, Week 4, No | 94 | 97 | 0
  Bloating, Week 5, Yes | 21 | 15 | 0
  Bloating, Week 5, No | 96 | 102 | 0
  Bloating, Week 6, Yes | 23 | 20 | 0
  Bloating, Week 6, No | 94 | 97 | 0
  Incomplete evacuation, Week 1, Yes | 16 | 10 | 17
  Incomplete evacuation, Week 1, No | 101 | 105 | 92
  Incomplete evacuation, Week 2, Yes | 23 | 14 | 24
  Incomplete evacuation, Week 2, No | 94 | 102 | 88
  Incomplete evacuation, Week 3, Yes | 20 | 18 | 21
  Incomplete evacuation, Week 3, No | 97 | 100 | 91
  Incomplete evacuation, Week 4, Yes | 21 | 18 | 0
  Incomplete evacuation, Week 4, No | 96 | 99 | 0
  Incomplete evacuation, Week 5, Yes | 24 | 20 | 0
  Incomplete evacuation, Week 5, No | 93 | 97 | 0
  Incomplete evacuation, Week 6, Yes | 24 | 20 | 0
  Incomplete evacuation, Week 6, No | 93 | 97 | 0
  Straining, Week 1, Yes | 21 | 8 | 14
  Straining, Week 1, No | 96 | 107 | 95
  Straining, Week 2, Yes | 21 | 17 | 19
  Straining, Week 2, No | 96 | 99 | 93
  Straining, Week 3, Yes | 19 | 23 | 21
  Straining, Week 3, No | 98 | 95 | 91
  Straining, Week 4, Yes | 22 | 21 | 0
  Straining, Week 4, No | 95 | 96 | 0
  Straining, Week 5, Yes | 25 | 22 | 0
  Straining, Week 5, No | 92 | 95 | 0
  Straining, Week 6, Yes | 21 | 21 | 0
  Straining, Week 6, No | 96 | 96 | 0
  IBS symptoms, Week 1, Yes | 29 | 22 | 30
  IBS symptoms, Week 1, No | 88 | 93 | 79
  IBS symptoms, Week 2, Yes | 42 | 22 | 30
  IBS symptoms, Week 2, No | 75 | 94 | 82
  IBS symptoms, Week 3, Yes | 37 | 30 | 29
  IBS symptoms, Week 3, No | 80 | 88 | 83
  IBS symptoms, Week 4, Yes | 37 | 33 | 0
  IBS symptoms, Week 4, No | 80 | 84 | 0
  IBS symptoms, Week 5, Yes | 35 | 30 | 0
  IBS symptoms, Week 5, No | 82 | 87 | 0
  IBS symptoms, Week 6, Yes | 41 | 29 | 0
  IBS symptoms, Week 6, No | 76 | 88 | 0

10. Secondary Outcome: Plasma Concentrations of GW876008 at Week 3 and 6
Description: For Week 3, 6, 9, 12, and 15 visits blood samples were collected at: pre-dose (after the pre ECG measurement and just before am dose) and immediately following the 1-3 hour post-dose ECG measurement and concentration of GW876008 was analyzed. Data for Week 3 and 6 was presented.
Time Frame: Week 3 and 6 visits. Pre-dose [after the pre Electrocardiogram (ECG) measurement and just before am dose] and immediately following the 1-3 hour post-dose ECG measurement
Population: Pharmacokinetic concentration population comprised of all participants for whom a pharmacokinetic sample was obtained and analyzed was included. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- GW876008 125 mg: Eligible participants received GW876008 125 mg once daily for 6 weeks Participants were instructed to take 1 tablet from each of the 2 bottles; 25 mg and 100 mg orally in the morning with food. At the day of the Weeks 3, 6, 9, 12 and 15 Visit, participants were instructed not take their dose prior to their visit which was scheduled for the morning, they were instructed to take their dose at the site after collection of a pre-dose PK blood sample.
Arm/Group | GW876008 125 mg
Number analyzed (Participants) | 107
ng/mL
  Week 3, pre dose | 672.691 (538.6495)
  Week 3, < 1 HR: number analyzed (Participants) | 1
  Week 3, < 1 HR | NA (NA) — Non Quantifiable
  Week 3, 1 to < 2 HR: number analyzed (Participants) | 93
  Week 3, 1 to < 2 HR | 1312.573 (716.2118)
  Week 3, 2 to < 3 HR: number analyzed (Participants) | 10
  Week 3, 2 to < 3 HR | 1170.096 (873.3578)
  Week 3, 3 to < 4 HR: number analyzed (Participants) | 3
  Week 3, 3 to < 4 HR | 966.653 (528.0190)
  Week 3, >= 4 HR: number analyzed (Participants) | 1
  Week 3, >= 4 HR | 696.690 (NA) — 1 participants was analyzed. thus S.D. was not calculated.
  Week 6, pre dose: number analyzed (Participants) | 99
  Week 6, pre dose | 625.645 (493.5978)
  Week 6, < 1 HR: number analyzed (Participants) | 6
  Week 6, < 1 HR | 850.028 (680.8931)
  Week 6, 1 to < 2 HR: number analyzed (Participants) | 84
  Week 6, 1 to < 2 HR | 1082.773 (656.4102)
  Week 6, 2 to < 3 HR: number analyzed (Participants) | 10
  Week 6, 2 to < 3 HR | 1004.535 (642.8820)

11. Secondary Outcome: IBS Composite Symptom Score
Description: Investigation of possible composite symptom score was planned. The data was not collected for composite symptom score.
Time Frame: Up to Day 105 (weeks 3-6 in period 1, weeks 12-15 in period 2)
Arm/Group | GW876008 125 mg | Placebo | Placebo Washout
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Changes in Patient Health Questionnaire-15 Somatization Scale (PHQ-15) Score With Treatment
Description: The PHQ-15 comprised of 15 somatic symptoms from the PHQ, each symptom scored from 0 to 2, where 0 ("Not bothered at all"), 1 (Bothered a little) 2 ("bothered a lot"). This questionnaire was completed at screening, and all study visits. Total score range was 0-30, where 0 indicated Not bothered at all and 30 indicated "bothered a lot". Higher score indicated greater severity of somatization symptoms.
Time Frame: Up to Day 105 (weeks 3-6 in period 1, weeks 12-15 in period 2)
Population: Intent to Treat population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | GW876008 125 mg | Placebo | Placebo Washout
Number analyzed (Participants) | 117 | 119 | 112
Score on a scale
  Week 3: number analyzed (Participants) | 111 | 115 | 112
  Week 3 | 8.6 (4.42) | 8.5 (3.89) | 8.5 (4.02)
  Week 6: number analyzed (Participants) | 105 | 113 | 0
  Week 6 | 8.8 (4.99) | 8.5 (4.03) |

13. Secondary Outcome: Summary of Anxiety and/or Depression on Hospital Anxiety and Depression Scale (HAD)
Description: HAD Scale was used to assess the severity of symptoms of anxiety and depression in participants. There were 14 questions. Seven questions related to depression and seven questions related to anxiety. Participants rated the severity of symptoms in the answer to each question. There were four options in each answer, from which participants had to select one. Responses were scored on a scale of 0, 1, 2 or 3, where 0 indicated best and 3 indicated worse. Total score ranged from 0-42 where 0 indicated absence of symptoms and higher scores indicated higher anxiety/depression complains. This questionnaire was completed at screening, and all study visits.
Time Frame: Up to Day 105 (weeks 3-6 in period 1, weeks 12-15 in period 2)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | GW876008 125 mg | Placebo | Placebo Washout
Number analyzed (Participants) | 112 | 117 | 111
Score on a scale
  Anxiety, Week 3 | 4.84 (3.690) | 4.68 (3.845) | 4.61 (3.749)
  Anxiety, Week 6: number analyzed (Participants) | 104 | 113 | 0
  Anxiety, Week 6 | 4.98 (4.141) | 4.56 (3.630) |
  Depression, Week 3: number analyzed (Participants) | 111 | 117 | 111
  Depression, Week 3 | 2.68 (3.027) | 2.79 (3.458) | 2.86 (3.297)
  Depression, Week 6: number analyzed (Participants) | 104 | 113 | 0
  Depression, Week 6 | 3.11 (3.612) | 2.50 (2.723) |

ADVERSE EVENTS:
Time Frame: Up to Day 147
Description: Safety population was used for AE,SAE and nSAE collection.
Arm/Group | GW876008 125 mg | Placebo | Placebo Washout
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/120 | 0/112
Serious Adverse Events (participants affected / at risk) | 0/119 | 1/120 | 0/112
Other Adverse Events (participants affected / at risk) | 9/119 | 5/120 | 2/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GW876008 125 mg (N=119) | Placebo (N=120) | Placebo Washout (N=112)
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GW876008 125 mg (N=119) | Placebo (N=120) | Placebo Washout (N=112)
Nasopharyngitis (Infections and infestations) | 9 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.